CLINICAL TRIAL: NCT05631288
Title: Association of Herpesvirus and Periodontitis: A Clinical and Laboratorial Case-control Study
Brief Title: Association of Herpesvirus and Periodontitis
Acronym: HerPerio
Status: Completed | Type: Observational
Sponsor: Miguel de Araújo Nobre (Other)
Collaborators: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor-Investigator, Miguel de Araújo Nobre, PhD, Malo Clinic
Organization: Malo Clinic (Other)
Other Study IDs: HerPerio
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Periodontitis
Keywords: periodontitis; herpes virus
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Unstimulated crevicular fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Periodontally compromised patients attending the Periodontology Department during periodontal diagnosis appointments at the point of first diagnosis.
  Interventions: Genetic: Sampe collection
- Controls: Periodontally healthy patients attending the remaining specialty departments ath the same clinic at the point of first diagnosis.
  Interventions: Genetic: Sampe collection

INTERVENTIONS:
Genetic: Sampe collection — Unstimulated crevicular fluid samples are collected using two sized 35 paper cones per subject, both used in the sampling process. The DNA is extracted from the samples through multiplex PCR at the Egas Moniz Applied Microbiology Laboratory (LMAEM).

SUMMARY:
A significant influence of the Herpes viruses family in the progression of periodontal disease has been suggested. The aim of this study was to investigate the potential association of four Herpes viruses (HSV-1, HSV-2, CMV and EBV) with periodontal disease using a qualitative test for evaluating the presence or absence of viral DNA in crevicular fluid samples of both healthy periodontal patients and periodontal compromised patients.

Adult patients with healthy periodontium or periodontally compromised attending the Egas Moniz university dental clinic (Almada, Portugal) are eligible to participate The study involves a periodontal diagnosis and collection of unstimulated crevicular fluid from saliva samples.

There will be no direct benefits for patients, but indirect benefit of advancing science in the study of potential involvment of Herpes viruses in periodontitis. No risks of participating are antecipated as the study material and data will be anonymized.

The study runs from the the Cooperativa de Ensino Egas Moniz and is expected to run for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients (> 18 years of age) with natural teeth attending clinical appointments at the Egas Moniz university dental clinic;
* Cases (periodontally compromised) included at the Department of Periodontology of the same clinic;
* Controls (periodontally healthy) included at the remaining departments of the same clinic.

Exclusion Criteria:

* Occurrence of a viral infection during the six months prior to the clinical study;
* Exposure to antiviral medication in the six months prior to the survey;
* Clinical history of immunosuppression, either exogenous or endogenous;
* Chemotherapy in the previous six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients (> 18 years of age) with natural teeth present attending clinical appointments at the Egas Moniz university dental clinic.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
The presence of virus DNA (HSV1, HSV2, EBV and CMV) | 1 day
  The presence of virus DNA (HSV1, HSV2, EBV and CMV)

SECONDARY OUTCOMES:
Smoking | one year
  [Smoking] (smoker, non-smoker) measured through questionnaire at first appointment;
Alcohol consumption | one year
  [Alcohol consumption] (yes, no) measured through questionnaire at first appointment;
Oral hygiene habits | one year
  [Oral hygiene habits] (0-1 times per day, 1-2 times per day and 2-3 times per day) measured through questionnaire at first time appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A de Araújo Nobre, PhD, Study Director — Maló Clinic
Locations (1):
- Malo Clinic, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
he datasets generated during and/or analysed during the current study will be available upon reasonable request.
Time Frame: 8 years
Access Criteria: Upon reasonable request